CLINICAL TRIAL: NCT00561080
Title: An Open-label, Randomised, Comparative, Multi-centre Study of the Immunogenicity and Safety of a 1-dose Regimen and Different 2-dose Regimens of a Zoster Vaccine (Live), ZOSTAVAX ®, in Subjects ≥ 70 Years of Age
Brief Title: Immunogenicity and Safety of a 1-dose Regimen of a Zoster Vaccine Versus Different 2-dose Regimens in Participants ≥ 70 Years of Age. (V211-043)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V211-043; X06-Z-305 (Other: MCMVaccBV (SPMSD) Protocol ID); 2007-000744-28 (EudraCT Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Prevention of : Herpes-Zoster
MeSH Terms: interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Single Dose of Zostavax (Experimental): Zostavax 0.65mL intramuscular injection administered on Day 0
  Interventions: Biological: Zostavax
- Zostavax - Day 0 and Month 1 (Experimental): Zostavax 0.65mL intramuscular injection administered on Day 0 and Month 1
  Interventions: Biological: Zostavax
- Zostavax - Day 0 and Month 3 (Experimental): Zostavax 0.65mL intramuscular injection administered on Day 0 and Month 3
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: Zostavax
  Other Names: Zoster vaccine live

SUMMARY:
Primary objective:

Immunogenicity To demonstrate that a second dose of ZOSTAVAX® elicits higher varicella-zoster virus (VZV) antibody titres than a first dose of ZOSTAVAX® whether given as a 0-1 month schedule or as a 0-3 month schedule in subjects ≥70 years of age as measured at 4 weeks post-vaccination

Secondary objectives Immunogenicity

* To summarise the VZV antibody titres at 4 weeks post-vaccination after a 1-dose regimen and 4 weeks post-vaccination after each dose of each 2-doses regimen of ZOSTAVAX®.
* To compare the VZV antibody titres at 12 months after completion of a 1-dose regimen with the VZV antibody titres at 12 months after completion of each 2-doses regimen of ZOSTAVAX®
* To summarise the VZV antibody titres at 24 and 36 months after completion of a 1-dose regimen and at 24 and 36 months after completion of each 2-doses regimen of ZOSTAVAX®

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years
2. Varicella history-positive or residence for > 30 years in a country with endemic VZV infection
3. Signed informed consent form prior to any study procedure

Exclusion Criteria:

1. Febrile illness within the last 72 hours before the first vaccination
2. Prior herpes-zoster episode clinically diagnosed by a physician
3. Prior receipt of varicella or zoster vaccine
4. Exposure to varicella or herpes-zoster within the 4 weeks prior to the first vaccination
5. Significant underlying illness preventing completion of the study vaccination schedules,
6. Known active tuberculosis,
7. Immune deficiency disorder, including active neoplastic disease within the prior 5 years,
8. Immune function impairment caused by medical condition or immunosuppressive therapy, or any other cause,
9. Receipt of any inactivated vaccine within the 2 weeks prior to the first vaccination,
10. Receipt of any other live vaccine within the 4 weeks prior to the first vaccination,
11. Receipt of immunoglobulins or blood-derived products within the 5 months prior to the first vaccination,
12. Concomitant use of non-topical antiviral therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 759 (Actual)
Dates: Start 2007-10-26 (Actual); Primary Completion 2009-06-03 (Actual); Study Completion 2009-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Vesikari T, Hardt R, Rumke HC, Icardi G, Montero J, Thomas S, Sadorge C, Fiquet A. Immunogenicity and safety of a live attenuated shingles (herpes zoster) vaccine (Zostavax(R)) in individuals aged >/= 70 years: a randomized study of a single dose vs. two different two-dose schedules. Hum Vaccin Immunother. 2013 Apr;9(4):858-64. doi: 10.4161/hv.23412. Epub 2013 Jan 14. PMID 23319176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 779 participants were screened. Twenty participants were not randomized.
Groups:
- Group 1: Single Dose of Zostavax: Single injection of the 0.65 mL of Zostavax administered on Day 0
- Group 2: Zostavax - Day 0 and Month 1: 0.65 mL of Zostavax administered on Day 0 and Month 1
- Group 3: Zostavax - Day 0 and Month 3: 0.65 mL of Zostavax administered on Day 0 and Month 3
Period: Vaccination Period (up to Month 4)
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Started | 253 | 255 | 251
Received at Least 1 Vaccination | 253 | 254 | 250
Completed | 250 | 229 | 225
Not Completed | 3 | 26 | 26
Not completed — Adverse Event | 0 | 4 | 6
Not completed — Definitive Contra-indication | 0 | 2 | 3
Not completed — Protocol Violation | 0 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 16 | 13
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 0 | 2 | 1
Period: 12-month Post Last Dose Follow-up
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Started | 250 | 229 | 225
Completed | 243 | 220 | 215
Not Completed | 7 | 9 | 10
Not completed — Adverse Event | 3 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 6 | 5
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: 24-month Post Last Dose Follow-up
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Started | 0 (Study stopped at 1 year post last dose) | 0 (Study stopped at 1 year post last dose) | 0 (Study stopped at 1 year post last dose)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0
Period: 36 Month Post Last Dose Follow-up
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Started | 0 (Study stopped at 1 year post last dose) | 0 (Study stopped at 1 year post last dose) | 0 (Study stopped at 1 year post last dose)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline age missing for 1 participant in Group 2 and 1 participant in Group 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3 | Total
Number analyzed (Participants) | 253 | 255 | 251 | 759
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline age missing for 1 participant in Group 2 and 1 participant in Group 3.
  years
    number analyzed (Participants) | 253 | 254 | 250 | 757
    (all) | 76.2 (5.5) | 76.0 (5.4) | 76.1 (5.3) | 76.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 138 | 135 | 421
  Male | 105 | 117 | 116 | 338

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Varicella Zoster Virus (VZV) Antibodies 4 Weeks After Each Vaccination: Groups 2 and 3
Description: Blood samples taken at 4 weeks post each vaccination to determine the geometric mean titer (GMT) of VZV antibodies via Glycoprotein Enzyme Linked Immunosorbent Assay (gpELISA).
Time Frame: 4 weeks post-dose 1 (Month 1 for all groups) and 4 weeks post-dose 2 (Month 2 for Group 2 and Month 4 for Group 3)
Population: All randomized participants in Groups 2 and 3 who received at least 1 dose of the study vaccine, had post-vaccination immunogenicity evaluation and excluded those with protocol violation which may have interfered with the immunogenicity evaluation or participants with herpes zoster (HZ) onset before the time point for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 203 | 198
gpELISA units/mL
  Post Dose 1 | 498.8 [438.7 to 567.1] | 523.3 [459.0 to 596.7]
  Post Dose 2 | 555.3 [496.6 to 620.9] | 410.5 [363.1 to 464.2]
Statistical Analysis 1: Comparison: Group 2: Zostavax - Day 0 and Month 1; Test type: Non-Inferiority or Equivalence — Superiority was achieved if the lower bound of the 2-sided 95% CI of the GMT ratio was greater than 1.2; p = 0.948, ANOVA; Geometric Mean Titer Ratio (GMTR) = 1.11, 95% CI 2-sided [1.02 to 1.22] — GMTR = GMT Post Dose 2/GMT Post dose 1
Statistical Analysis 2: Comparison: Group 3: Zostavax - Day 0 and Month 3; Test type: Non-Inferiority or Equivalence — Superiority was achieved if the lower bound of the 2-sided 95% CI of the GMT ratio was greater than 1.2; p > 0.999, ANOVA; GMTR = 0.78, 95% CI 2-sided [0.73 to 0.85] — GMTR = GMT Post Dose 2/GMT Post dose 1

2. Secondary Outcome: Geometric Mean Titer (GMT) of VZV Antibodies 4 Weeks After Vaccination: Group 1
Description: Blood sample taken at 4 weeks post vaccination to determine the geometric mean titer (GMT) of VZV antibodies via gpELISA.
Time Frame: 4 weeks post-dose (Month 1)
Population: All randomized participants in Group 1 who received study vaccine, had post-vaccination immunogenicity evaluation and excluded those with protocol violation which may have interfered with the immunogenicity evaluation or participants with herpes zoster (HZ) onset before the time point for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Group 1: Single Dose of Zostavax
Number analyzed (Participants) | 243
gpELISA units/mL
  GMT Pre-Dose: number analyzed (Participants) | 242
  GMT Pre-Dose | 233.7 [207.1 to 263.7]
  GMT Post Dose | 550.0 [489.2 to 618.4]
Statistical Analysis 1: Comparison: Group 1: Single Dose of Zostavax; Test type: Superiority or Other; GMFR = 2.35, 95% CI 2-sided [2.11 to 2.62] — GMFR=GMT Post Dose/GMT Pre Dose

3. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titres From Pre-vaccination to 4 Weeks Post-dose 1 in Groups 1, 2 and 3 and 4 Weeks Post-dose 2 in Groups 2 and 3
Description: Blood sample taken at predose (Day 0) and 4 weeks post each vaccination to determine the geometric mean titer (GMT) of VZV antibodies via gpELISA. The GMFR was calculated following each vaccination as GMT Post-dose/GMT Pre-vaccination
Time Frame: Predose and 4 weeks post-dose 1 (Month 1 for all groups) and 4 weeks post-dose 2 (Month 2 for Group 2 and Month 4 for Group 3)
Population: All randomized participants in who received at least 1 dose of the study vaccine, had pre-dose 1 evaluation and had post-vaccination immunogenicity evaluation. Excluded those with protocol violation which may have interfered with the immunogenicity evaluation or participants with herpes zoster (HZ) onset before the time point for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 242 | 203 | 198
gpELISA units/mL
  GMFR Post Dose 1 | 2.35 [2.11 to 2.62] | 2.37 [2.11 to 2.66] | 2.29 [2.05 to 2.57]
  GMFR Post Dose 2 | NA [NA to NA] — Group 1 did not have 2nd vaccination | 2.64 [2.37 to 2.95] | 1.80 [1.63 to 1.98]

4. Secondary Outcome: Geometric Mean Titre of VZV Antibodies 12 Months Post-last Dose
Description: Blood sample taken at 1 year post last vaccination to determine the geometric mean titer (GMT) of varicella antibodies via gpELISA.
Time Frame: 1 year post final dose for Groups 1, 2, and 3 (Group 1: Month 12; Group 2: 13 Month 13; and Group 3: Month 15)
Population: All randomized participants in who received at least 1 dose of the study vaccine, had 12-month post-vaccination immunogenicity evaluation and excluded those with protocol violation which may have interfered with the immunogenicity evaluation or participants with herpes zoster (HZ) onset before the time point for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 223 | 189 | 204
gpELISA units/mL | 246.8 [230.9 to 263.9] | 261.1 [242.8 to 280.7] | 266.6 [248.6 to 285.8]
Statistical Analysis 1: Comparison: Group 1: Single Dose of Zostavax vs Group 2: Zostavax - Day 0 and Month 1; ANCOVA model includes country and age at first vaccination as independent variables and baseline antibody titre as covariate. The GMT 12-month post-last dose is the GMT adjusted from the ANCOVA model; Test type: Superiority or Other; GMT Ratio = 1.06, 95% CI 2-sided [0.96 to 1.17] — GMT Ratio = Group 2 GMT/Group 1 GMT
Statistical Analysis 2: Comparison: Group 1: Single Dose of Zostavax vs Group 3: Zostavax - Day 0 and Month 3; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; GMT Ratio = 1.08, 95% CI 2-sided [0.98 to 1.19] — GMT Ratio = GMT Group 3/GMT Group 1

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titres From Pre-Vaccination To 12 Months Post-dose 1 in Group 1 And From Pre-Vaccination To 12 Months Post-dose 2 in Groups 2 and 3
Description: Blood sample taken at predose and 1 year post last vaccination to determine the GMFR of varicella antibodies via gpELISA. Geometric mean fold rise was calculated for each arm as GMT 12-month post last dose divided by pre-vaccination GMT.
Time Frame: predose 1 and 1 year post-last dose (Group 1: Month 12; Group 2: 13 Month 13; and Group 3: Month 15)
Population: All randomized participants who received at least 1 dose of the study vaccine, had 12-month post-vaccination immunogenicity evaluation and excluded those with protocol violation which may have interfered with the immunogenicity evaluation or participants with herpes zoster (HZ) onset before the time point for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 223 | 189 | 204
gpELISA units/mL | 1.06 [0.99 to 1.14] | 1.16 [1.06 to 1.26] | 1.17 [1.07 to 1.27]

6. Secondary Outcome: Geometric Mean Titre (GMT) of VZV Antibodies 24 and 36 Months Post-dose 1 in Group 1 and the 24 and 36 Months Post-dose 2 in Groups 2 and 3
Description: Blood sample taken at 36 months post last-vaccination to determine the geometric mean titer (GMT) of varicella antibodies via gpELISA.
Time Frame: 24 and 36 months post-last dose
Population: Study stopped after 12 months. As per protocol, the study was stopped after the 12-month follow-up since there was no statistical evidence or clinical trend for superiority of any of the 2-dose regimens compared with the 1-dose regimen. 24 and 36 month data not obtained.
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titres From Pre-Vaccination To 24 And 36 Months Post-dose 1 in Group 1 and From Pre-vaccination To 24 And 36 Months Post-dose 2 in Groups 2 and 3
Description: Blood samples were to be taken at predose and 24 months post- last vaccination in Groups 1 , 2, and 3 to determine the GMFR of varicella antibodies via gpELISA. Geometric mean fold rise was to be calculated for each arm as GMT 24-month post last dose divided by pre-vaccination GMT.
Time Frame: Predose 1 and 24 and 36 months post-last dose
Population: as for outcome 6
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Reported a Solicited Injection Site Reaction : Post-dose 1
Description: Participants entered data into daily dairy card regarding previously identified possible injection site reactions of erythema, injection site swelling or injection site pain
Time Frame: up to 4 days after 1st vaccination
Population: All randomized participants in Groups 1, 2 and 3 who received the 1st dose of study drug and had follow-up safety data. .
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 47.2 | 46.0 | 42.2

9. Secondary Outcome: Percentage of Participants Who Reported a Solicited Injection Site Reaction: Post-dose 2
Description: as for outcome 8
Time Frame: up to 4 days after 2nd vaccination
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 42.2 | 42.1

10. Secondary Outcome: Percentage of Participants Who Reported an Unsolicited Injection Site Reaction: Post-dose 1
Description: The percentage of participants who reported an injection site reaction that was not specifically prompted by the diary card within 28 day of 1st vaccination was recorded.
Time Frame: up to 28 days after 1st of study drug
Population: All randomized participants in Groups 1, 2, and 3 who received at least 1 dose of study drug and had follow-up safety data. .
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 5.6 | 4.8 | 0.8

11. Secondary Outcome: Percentage of Participants Who Reported an Unsolicited Injection Site Reaction: Post-dose 2
Description: The percentage of participants that reported an injection site reaction that was not specifically prompted by the diary card within 28 days post-dose 2 was recorded.
Time Frame: up to 28 days post-dose 2
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of study drug and had follow-up safety data. .
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 1.3 | 3.2

12. Secondary Outcome: Percentage of Participants Who Reported Herpes Zoster or Zoster-like Rash: Post-dose 1
Description: Percentage of participants who reported herpes zoster or zoster-like rash following the 1st dose of vaccine were recorded.
Time Frame: up to 28 days post-dose 1
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of the study drug and who have safety follow-up data for post-dose 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 0.8 | 0.0 | 0.0

13. Secondary Outcome: Percentage of Participants Who Reported Herpes Zoster or Zoster-like Rash: Post-Dose 2
Description: Percentage of participants who reported herpes zoster or zoster-like rash following the 2nd dose of vaccine were recorded.
Time Frame: up to 28 days post-dose 2
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of the study drug and who have safety follow-up data for post-dose 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 0.0 | 0.0

14. Secondary Outcome: Percentage of Participants Who Reported Varicella or Varicella-like Rash: Post-dose 1
Description: Percentage of participants that reported varicella or varicella-like rash following the 1st dose of vaccine were recorded.
Time Frame: up to 28 days post-dose 1
Population: All randomized participants in Groups 1, 2 and 3 who received 1st dose of the study drug and who have safety follow-up data for post-dose 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 0.0 | 0.0 | 0.0

15. Secondary Outcome: Percentage of Participants Who Reported Varicella or Varicella-like Rash: Post-dose 2
Description: Percentage of participants that reported varicella or varicella-like rash following the 2nd dose of vaccine were recorded.
Time Frame: up to 28 days post-dose 2
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 0.4 | 0.5

16. Secondary Outcome: Percentage of Participants Who Reported a Systemic Adverse Event: Post-dose 1
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Adverse events that were considered systemic (not localized) were summarized
Time Frame: up to 28 days after 1st vaccination
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of study drug and had follow-up safety data. .
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 25.8 | 32.7 | 25.7

17. Secondary Outcome: Percentage of Participants Who Reported a Systemic Adverse Event: Post-dose 2
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Adverse events that were considered systemic (not localized) were summarized,
Time Frame: up to 28 days after 2nd vaccination
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 20.7 | 15.4

18. Secondary Outcome: Percentage of Participants Who Reported a Vaccine-related Systemic Adverse Event: Post-dose 1
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Adverse events that were considered systemic (not localized) and were reported as at least possibly related to the vaccine were summarized
Time Frame: up to 28 days after 1st vaccination
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of study drug and had follow-up safety data. .
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 6.7 | 4.0 | 8.4

19. Secondary Outcome: Percentage of Participants Who Reported a Vaccine-related Systemic Adverse Event: Post-dose 2
Description: An adverse event (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Adverse events that were considered systemic (not localized) and were reported as at least possibly related to the vaccine were summarized,
Time Frame: up to 28 days after 2nd vaccination
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 3.4 | 2.7

20. Secondary Outcome: Percentage of Participants Who Reported a Serious Adverse Event: Post-dose 1
Description: A serious adverse event (SAE) is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement. The percentage of participants who reported an SAE within 28 days of 1st dose of vaccine were recorded.
Time Frame: up to 28 days after 1st vaccination
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 0.4 | 2.8 | 0.4

21. Secondary Outcome: Percentage of Participants Who Reported a Serious Adverse Event: Post-dose 2
Description: as for outcome 20
Time Frame: up to 28 days after 2nd vaccination
Population: All randomized participants in Groups 2 and 3 who received 2nd dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 0 | 232 | 221
Percentage of Participants |  | 0.9 | 0.9

22. Secondary Outcome: Percentage of Participants Who Reported a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement. The percentage of participants who reported an SAE during the entire study period that was considered at least possibly -related to the vaccine were recorded.
Time Frame: up to end of study (approximately 15 months)
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Percentage of Participants Who Died During the Study
Description: The number of participants who died for any reason during the study was summarized.
Time Frame: up to end of study (approximately 15 months)
Population: All randomized participants in Groups 1, 2, and 3 who received 1st dose of study drug and had follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Number analyzed (Participants) | 252 | 248 | 249
Percentage of Participants | 1.6 | 2.0 | 1.2

ADVERSE EVENTS:
Time Frame: up to 1 year post-last dose (Group 1: 12 months total; Group 2: 13 months total; Group 3: 14 months total)
Description: Analysis population is all enrolled participants.
Arm/Group | Group 1: Single Dose of Zostavax | Group 2: Zostavax - Day 0 and Month 1 | Group 3: Zostavax - Day 0 and Month 3
Serious Adverse Events (participants affected / at risk) | 4/253 | 11/255 | 4/251
Other Adverse Events (participants affected / at risk) | 122/253 | 144/255 | 132/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Single Dose of Zostavax (N=253) | Group 2: Zostavax - Day 0 and Month 1 (N=255) | Group 3: Zostavax - Day 0 and Month 3 (N=251)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Single Dose of Zostavax (N=253) | Group 2: Zostavax - Day 0 and Month 1 (N=255) | Group 3: Zostavax - Day 0 and Month 3 (N=251)
Injection site erythema (General disorders) | 107 (107) | 125 (185) | 122 (181)
Injection site pain (General disorders) | 57 (60) | 75 (98) | 74 (101)
Injection site swelling (General disorders) | 69 (69) | 73 (106) | 67 (92)
Headache (Nervous system disorders) | 13 (16) | 14 (18) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must first obtain written consent from Sanofi Pasteur MSD. If consent is given, all abstracts manuscripts, texts, or presentation, etc... shall be sent to Sanofi Pasteur MSD for review and approval prior to their publication or presentation. Sanofi Pasteur MSD shall have sixty days to review these documents and may refuse to give its consent in part or whole for confidential reasons (including but not limited to intellectual property rights, whether patentable or not).